CLINICAL TRIAL: NCT07124715
Title: Dynamic Navigation for Zygomatic Implant Rehabilitation: An Innovative Protocol Using an Intraoral Reference System and Evaluation of a New Zygomatic Implant Design
Brief Title: Dynamic Navigation for Zygomatic Implant Rehabilitation Using an Intraoral Reference System: Evaluation of a New Zygomatic Implant Design
Acronym: NAVIZYG-SURF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Pietro Felice, Principal Investigator, Head of Oral Surgery, Clinical Professor, University of Bologna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ZYGOMA01.17
Record Dates: First submitted 2025-07-31; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Atrophic Maxilla; Zygomatic Implants; Implant Surface
Keywords: bone loss; zygomatic implants; implant surface; atrophic maxilla; oral rehabilitation; perimplantitis
MeSH Terms: conditions — Atrophic Maxilla; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Rough Surface Zygomatic Implant (Active Comparator): Patients receive a zygomatic implant with a fully roughened surface (from apex to collar) on one side of the maxilla. Implant placement is performed using dynamic navigation. This arm serves as the control in a split-mouth randomized design.
  Interventions: Device: Rough Surface Zygomatic Implant
- Modified Partially Machined Surface Zygomatic Implant (Experimental): Patients receive a zygomatic implant with a modified surface, including a smooth machined coronal portion, a non-threaded machined intermediate section, and a rough apical portion, on the contralateral side of the maxilla. Implant placement is performed using dynamic navigation. This arm represents the test condition in the split-mouth design.
  Interventions: Device: Partially Machined Surface Zygomatic Implant

INTERVENTIONS:
Device: Rough Surface Zygomatic Implant — Surgical placement of a zygomatic implant with a fully roughened surface from apex to collar. Used for the control arm.
  Arms: Standard Rough Surface Zygomatic Implant
Device: Partially Machined Surface Zygomatic Implant — Surgical placement of a modified zygomatic implant with a smooth machined coronal portion, a non-threaded machined middle section, and a rough apical portion. Used for the test arm.
  Arms: Modified Partially Machined Surface Zygomatic Implant

SUMMARY:
This clinical study aims to evaluate the effectiveness and safety of zygomatic implants placed using dynamic navigation technology. Specifically, it compares two types of zygomatic implants with different surface characteristics: one with a fully rough surface and another with a partially smooth (machined) surface near the gum line. The goal is to determine whether surface design affects surgical performance, healing, implant success, and patient outcomes. A total of 22 patients with severe upper jaw bone loss will receive both types of implants-one on each side of the upper jaw-in a randomized, split-mouth design. The study also evaluates pain, swelling, healing time, and patient quality of life over a 5-year follow-up period.

DETAILED DESCRIPTION:
This prospective, randomized, split-mouth clinical study investigates the use of dynamic navigation for the placement of zygomatic implants in patients with severely atrophic maxillae. The primary aim is to compare two different surface configurations of zygomatic implants: a fully rough surface versus a partially machined (smooth) coronal surface. Each of the 22 enrolled patients will receive both implant types-one per side-allowing for direct intra-patient comparison.

All surgeries are planned using three-dimensional imaging and performed with a dynamic navigation system (ImplaNav), calibrated for the longer drills required for zygomatic implant sites. The study evaluates surgical accuracy, implant stability, preparation time, postoperative pain and swelling, sinus membrane response, and long-term implant and prosthetic success. Patient quality of life is also monitored over a 5-year follow-up using standardized questionnaires and radiographic assessments.

This study aims to provide evidence on whether implant surface design influences clinical performance and healing outcomes in zygomatic implant rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Patients requiring partial or full rehabilitation of the atrophic maxilla

Candidates for placement of at least one zygomatic implant per side (right and left), connected to at least one standard or zygomatic implant

Severe maxillary atrophy confirmed by CT scan, with insufficient bone for conventional implants or only sufficient bone for 2 frontal implants (minimum diameter 3.5 mm, length 8 mm)

Residual alveolar crest height ≤ 4 mm beneath the maxillary sinus

Age ≥ 18 years

Signed informed consent

Exclusion Criteria:

General contraindications to oral surgery

History of radiation therapy to the head and neck exceeding 70 Gy

Compromised or suppressed immune system

Current or past use of intravenous bisphosphonates

Uncontrolled diabetes mellitus

Alcohol or drug dependency

Psychiatric disorders

Pregnancy or breastfeeding

Participation in other clinical trials

Inability to attend a 5-year follow-up

Limited mouth opening (< 3.5 cm interincisal distance)

Absence of opposing dentition or lower prosthesis

Acute or chronic infection in the intended implant site

Untreated active periodontal disease

Poor oral hygiene motivation

Radiographic signs of sinus membrane inflammation or ostium obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Implant Success Rate of Zygomatic Fixtures | 5 years after implant placement
  The success of each zygomatic implant will be assessed clinically by evaluating the absence of pain, absence of mobility or rotation under contra-torque testing, and the presence of healthy peri-implant tissues. Clinical evaluation will be supported by radiographic analysis to confirm peri-implant bone maintenance and the absence of pathological signs.

SECONDARY OUTCOMES:
Surgical Site Preparation Time | Intraoperative (during implant placement)
  Time required to prepare each zygomatic implant site will be recorded, from the start of the first drill to the complete insertion of the implant. The comparison aims to detect differences between the rough and partially machined implant groups.
Radiographic Evaluation of Peri-Implant Bone | At prosthesis delivery, and at 1, 3, and 5 years post-loading
  Assessment of peri-implant bone levels will be performed through standardized radiographs (OPT and teleradiography) and analyzed using calibrated software. Bone changes will be compared between implant types.
Peri-implant Probing Depth (PD) | 1, 3, and 5 years after functional loading
  Mean probing depth, in millimetres, measured circumferentially around each implant to assess peri-implant soft-tissue health. Results will be reported as mean ± SD per implant.
Number of Implants with Bleeding on Probing (BOP) | 1, 3, and 5 years after functional loading
  Count of dental implants that exhibit bleeding upon gentle circumferential probing (≤ 0.25 N). The result will be reported as the total number of affected implants and the corresponding percentage of all implants examined at each follow-up visit.
Number of Implants with Suppuration | 1, 3, and 5 years after functional loading
  Count of dental implants showing the presence of suppuration (pus discharge) upon gentle probing (≤ 0.25 N) during clinical examination. The result will be reported as the number and percentage of affected implants at each follow-up visit.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung K, Huang W, Wang F, Wu Y. Real-Time Surgical Navigation System for the Placement of Zygomatic Implants with Severe Bone Deficiency. Int J Oral Maxillofac Implants. 2016 Nov/Dec;31(6):1444-1449. doi: 10.11607/jomi.5526. PMID 27861671
- [Background] Branemark PI, Grondahl K, Ohrnell LO, Nilsson P, Petruson B, Svensson B, Engstrand P, Nannmark U. Zygoma fixture in the management of advanced atrophy of the maxilla: technique and long-term results. Scand J Plast Reconstr Surg Hand Surg. 2004;38(2):70-85. doi: 10.1080/02844310310023918. PMID 15202664
- [Background] Esposito M, Grusovin MG, Felice P, Karatzopoulos G, Worthington HV, Coulthard P. Interventions for replacing missing teeth: horizontal and vertical bone augmentation techniques for dental implant treatment. Cochrane Database Syst Rev. 2009 Oct 7;2009(4):CD003607. doi: 10.1002/14651858.CD003607.pub4. PMID 19821311
- [Background] Branemark PI, Hansson BO, Adell R, Breine U, Lindstrom J, Hallen O, Ohman A. Osseointegrated implants in the treatment of the edentulous jaw. Experience from a 10-year period. Scand J Plast Reconstr Surg Suppl. 1977;16:1-132. No abstract available. PMID 356184